CLINICAL TRIAL: NCT01527929
Title: An Open-label Pharmacokinetic and Safety Study of Cabazitaxel in Patients With Solid Tumors With Moderately and Severely Impaired and With Normal Renal Function
Brief Title: Pharmacokinetics and Safety Study of Cabazitaxel in Cancer Patients With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POP12251; 2011-001517-14 (EudraCT Number); U1111-1121-4512 (Other: UTN)
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A (Experimental): Normal renal function - Cabazitaxel administered once every 3 weeks
  Interventions: Drug: Cabazitaxel XRP6258
- Cohort B (Experimental): Moderate renal dysfunction - Cabazitaxel administered once every 3 weeks
  Interventions: Drug: Cabazitaxel XRP6258
- Cohort C (Experimental): Severe renal dysfunction - Cabazitaxel administered once every 3 weeks
  Interventions: Drug: Cabazitaxel XRP6258

INTERVENTIONS:
Drug: Cabazitaxel XRP6258 — Pharmaceutical form: solution for infusion Route of administration: intravenous

SUMMARY:
Primary Objective:

- To assess potential impact of moderate and severe renal impairment on the pharmacokinetics of cabazitaxel

Secondary Objective:

- To assess the safety of cabazitaxel in patients with various degrees of renal impairment

DETAILED DESCRIPTION:
The study consists of a screening phase, registration, cabazitaxel administration will start within 5 business days of registration, with 21-day study treatment cycles. Cycle lengths may be extended up to a maximum of 14 additional days in case of unresolved toxicity. Patients continue to receive treatment until they experience, unacceptable toxicities/Adverse Events, disease progression, withdraw their consent, or the investigator decides to discontinue the patient, and the subsequent 30 days follow-up or study cut-off, whichever comes first.

Patients may continue to be treated as long as they are benefiting from study treatment and have not met study withdrawn criteria.

ELIGIBILITY:
Inclusion criteria :

* Diagnosis of histologically or cytologically proven non-hematologic malignancy. The cancer must be one that is either refractory to standard therapy or for which no standard therapy exists. Cabazitaxel is an adequate treatment option, as judged by investigator.
* Eastern Cooperative Oncology Group performance status 0 - 2
* Stable renal function
* Patients must have adequate liver and marrow function as defined below:

  * Absolute neutrophil count ≥ 1.5x10^9/L
  * Platelets ≥ 100x10^9/L
  * Total bilirubin ≤ 1.0 x the institutions upper limit of normal
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 x the institutions upper limit of normal
  * Alkaline phosphatase ≤ 2.5 x the institutions upper limit of normal
* Patient may have a Grade 1 or less neurotoxicity at study entry.
* Life expectancy > 3 months
* Age ≥ 18 years old
* If female, subject must use a double contraception method, except if she is sterilized for more than 3 months or postmenopausal.
* Having given written informed consent prior to any procedure related to the study

Exclusion criteria:

* Less than 4 weeks have elapsed from prior anticancer therapy (surgery, chemotherapy, radiation therapy, hormonal therapy and immunotherapy). Prior isotope therapy and radiotherapy to ≥ 30% of bone marrow are not allowed.
* Any of the following within 6 months prior to study enrollment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, class III or IV congestive heart failure, stroke or transient ischemic attack.
* Any of the following within 3 months prior to study start: treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism, or other uncontrolled thromboembolic event.
* Active hepatitis
* Acute renal failure (new or superimposed to pre-existing chronic renal impairment), nephrotic syndrome.
* Patients requiring dialysis during the study.
* History of hypersensitivity to docetaxel or polysorbate 80.
* Known acquired immunodeficiency syndrome (AIDS-related illnesses) or known HIV disease requiring antiretroviral treatment.
* Known brain metastases.
* If female, pregnancy or breast-feeding.
* Any treatment known to induce CYP isoenzymes (e.g., phenobarbital, phenytoin, carbamazepine, rifampicin, St John's Wort) or to strongly inhibit CYP3A4 activities (e.g., ketoconazole, itraconazole, macrolides, antiprotease agents, etc) is not allowed within 2 weeks before or during the test period of the pharmacokinetic sampling

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of cabazitaxel in study population | Up to day 10

SECONDARY OUTCOMES:
Safety profile of cabazitaxel in study population, as measured by adverse events, clinical, laboratory and ECG parameters | up to 30 days after the last dosing

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Belgium (2):
  - Investigational Site Number 056002, Brussels
  - Investigational Site Number 056001, Ghent
- Investigational Site Number 380001, Milan, Italy
- Netherlands (2):
  - Investigational Site Number 528001, Rotterdam
  - Investigational Site Number 528002, Utrecht
- Investigational Site Number 724001, Barcelona, Spain
- Investigational Site Number 826001, Cambridge, United Kingdom